CLINICAL TRIAL: NCT01322152
Title: Phase II Study of Irinotecan Plus Capecitabine as the First-line or Second-line Treatment for Advanced Colorectal Cancer Patients
Brief Title: Study of Irinotecan Plus Capecitabine to Treat Advanced Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jin Li, Dr, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XELIRIcrc
Record Dates: First submitted 2011-03-23; First posted 2011-03-24 (Estimated); Last update posted 2013-06-11 (Estimated); Status verified 2013-06

CONDITIONS: Colorectal Cancer
Keywords: metastases; neoplasm
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Neoplasms | interventions — Irinotecan; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- wXELIRI regimen (Experimental)
  Interventions: Drug: irinotecan, capecitabine

INTERVENTIONS:
Drug: irinotecan, capecitabine — Irinotecan: 90 mg/m2, d1, iv gtt; Capecitabine: 1200mg/m2 Bid, d1-5, po; The regimen is repeated every 7 days.

SUMMARY:
The objectives of this study are to evaluate the efficacy and tolerability of single-week regimen of irinotecan plus capecitabine in the first-line or second-line treatment of advanced colorectal cancer.

DETAILED DESCRIPTION:
Irinotecan and capecitabine are approved to be the effective drugs for the advanced colorectal cancer patients. However, the combination of these two drugs are not regularly recommended due to the severe diarrhea as the most common adverse event.This study was designed to explore whether the single-week regimen of irinotecan plus capecitabine improves efficacy and does not increase the toxicity in advanced colorectal cancer patients in China.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Histologically confirmed colorectal cancer
* Age 18-70 years old
* Advanced colorectal cancer patients, first-line or second-line treatment, the adjuvant treatment including the oxaliplatin or/and 5FU should be finished six months before
* Have at least one measurable lesion according to the Response Evaluation Criteria in Solid Tumors (RECIST) criteria.
* ECOG 0-1
* Life expectancy of more than 3 months.
* Normal laboratory values: hemoglobin > 90g/dl, neutrophils > 1.5×10^9/L, platelets > 100×10^9/L, serum creatinine < 1.5×upper limit of normal (ULN), serum bilirubin < 1.5×ULN, ALT and AST < 2.5×ULN, AKP < 4×ULN

Exclusion Criteria:

* Pregnant or lactating patients
* Concurrent disease or condition that would make the subject inappropriate for study participation, or any serious medical disorder that would interfere with the subject's safety
* Active or uncontrolled infection
* Known history of uncontrolled or symptomatic angina, arrhythmias, or congestive heart failure
* Patients could not swallow the tablets
* Concomitant with brain metastases

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2011-03; Primary Completion 2013-05 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Rate of Diarrhea | eight weeks

SECONDARY OUTCOMES:
Progression free survival | eight weeks
Response rate | eight weeks
Disease control rate | eight weeks
Overall survival | eight weeks
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | eight weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, PhD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Li W, Xu J, Shen L, Liu T, Guo W, Zhang W, Chen Z, Zhu X, Li J. Phase II study of weekly irinotecan and capecitabine treatment in metastatic colorectal cancer patients. BMC Cancer. 2014 Dec 19;14:986. doi: 10.1186/1471-2407-14-986. PMID 25527007